CLINICAL TRIAL: NCT07301788
Title: A Mechanistic Study on the Impact of Donor Heart Procurement Time on Recipient Prognosis After Heart Transplantation Based on Multi-Omics Analysis
Brief Title: Donor Circadian Rhythm and Its Correlation With Prognosis After Heart Transplantation
Acronym: CIRCA-HTx
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0291; JCZRYB202500142 (Other Grant/Funding Number: Hubei Provincial Natural Science Foundation Projects); 2021YFA1101900 (Other Grant/Funding Number: National Key Research and Development Program); 82470423 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Heart Transplantation; End-stage Heart Failure; Circadian Rhythm
Keywords: Heart transplant; Donor heart procurement; Circadian Rhythm; Transplant outcomes; Survival analysis; Rejection; End-stage heart failure; Biomarkers; Multi-omics; Observational study; Prognostic factors
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Donor left atrial appendages of surgical waste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the impact of donor heart procurement time based on circadian rhythm on the long-term outcomes of heart transplant recipients. The main question it aims to answer is:

Does the time of day when a donor heart is procured-specifically during the circadian repression phase (00:00-12:00) versus the activation phase (12:00-00:00)-affect post-transplant survival and rejection rates in patients with end-stage heart failure?

Patients undergoing heart transplantation at the study hospital will have leftover donor heart tissue and preservation fluid collected during surgery for multi-omics analysis. These participants will then be followed prospectively for up to three years to track survival and rejection outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing heart transplantation surgery at our hospital due to end-stage heart failure.

Exclusion Criteria:

* Exclude patients undergoing multi-organ combined transplantation, re-do heart transplantation, or those with a history of other organ transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients diagnosed with end-stage heart failure who are scheduled to undergo heart transplantation at the study hospital. Participants must meet standard transplant eligibility criteria. Exclusion criteria are applied to minimize confounding factors, including previous organ transplants, re-transplants, and multi-organ transplant recipients, ensuring a more homogeneous study population focused on first-time, heart-only transplant cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of transplantation up to 3 years post-transplant.
  Post-heart-transplant survival assessed from the date of transplantation until death from any cause, evaluated through regular follow-up visits over the study period.

SECONDARY OUTCOMES:
Acute rejection rate | From date of transplantation up to 3 years post-transplant.
  Incidence of acute cellular rejection following heart transplantation, diagnosed based on endomyocardial biopsy per International Society of Heart and Lung Transplantation (ISHLT) grading criteria (grade 2R or higher).

CONTACTS AND LOCATIONS:
Overall Officials: Nianguo Dong, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared publicly. All data collected will be used solely by the research team for the analysis purposes outlined in this protocol.